CLINICAL TRIAL: NCT01679964
Title: A Single Arm Study to Assess the Sustained Virological Suppression and Improvement of Treatment-emerged Adverse Events of Switching to Raltegravir in Stable HIV-infected Patients on Ritonavir-boosted Protease Inhibitor Regimen
Brief Title: Sustained Virological Suppression and Improvement of Adverse Events of Switching to Raltegravir Study
Acronym: TaISENWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lin, Hsi-Hsun, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISP40301; MISP 40301 (Other Grant/Funding Number: MISP 40301)
Record Dates: First submitted 2012-08-30; First posted 2012-09-06 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: HIV Infection; Adverse Drug Reaction; Quality of Life
Keywords: HIV infection; Raltegravir; Adverse event; Life quality
MeSH Terms: conditions — HIV Infections; Drug-Related Side Effects and Adverse Reactions | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir switch (Other): Isentress (400mg) bid + 2 NRTI (at least 2 nucleoside or nucleotide reverse transcriptase inhibitors and no other protease inhibitors)
  Interventions: Drug: Raltegravir switch

INTERVENTIONS:
Drug: Raltegravir switch — Isentress (400mg) bid + 2 NRTI (at least 2 nucleoside or nucleotide reverse transcriptase inhibitors and no other protease inhibitors)
  Other Names: Isentress

SUMMARY:
Switching from the ritonavir-boosted protease inhibitor component to raltegravir in stable HIV-infected adult patients receiving combination therapy will demonstrate improved clinical tolerability or lipid profiles with sustained plasma virological response (<50 copies/ml).

DETAILED DESCRIPTION:
A. Objectives To compare the treatment-emerged AEs and virological suppression after switch to raltegravir-based therapy in stable HIV-infected patients who receiving ritonavir-boosted protease inhibitor antiretroviral regimen

Primary endpoints:

1) The changes in overall incidence and severity of patient-reported clinical adverse events (based on "symptom distress module) after switch to raltegravir-based therapy.

Secondary endpoints:

1. The proportion of patients who are free of "virological failure" at week 48 after switch
2. The change from baseline in CD4 cell counts at week 48 after switch
3. The change in quality of life by assess the changes in the domain scores of MOS-HIV questionnaire at baseline and different study time points.
4. The changes in laboratory adverse event, e.g., the mean percent changes from baseline to 48 weeks in plasma lipid profile (total cholesterol, LDLCholesterol, HDL Cholesterol, triglycerides) after switch
5. The proportion of patients who are free of "treatment failure" at week 48 after switch

Safety endpoints

1. Incidence of adverse events
2. The proportion of patients with treatment-related grade 3 or 4 adverse events and laboratory abnormalities

ELIGIBILITY:
Inclusion Criteria:

* Patients who are infected with HIV-1
* Ages at least 20 years
* Patients are currently receiving a ritonavir-boosted PI-based regimen, including lopinavir, atazanavir, or darunavir, plus at least 2 antiretroviral agents (NRTIs)
* Patient complained of treatment-emerged clinical adverse events or abnormal lipid profile
* Patients with plasma HIV-1 viral RNA below 50 copies per ml for at least 6 months

Exclusion Criteria:

* Patient with known history of contraindication or hypersensitivity to any component of the study regimen
* Patients with acute or decompensated chronic hepatitis in the previous 6 months
* Patients with chronic hepatitis and serum aminotransferase concentrations are more than 5 times the upper limit of the normal range
* Patients with renal insufficiency (patients need dialysis or have serum creatinine concentrations of more than twice the upper limit of the normal range
* Current alcohol or substance abuse (patients receiving methadone for the management of withdrawal symptoms due to substance abuse are allowed )
* Patients have failed previous regimens (prior to starting the current 2NRTI+PI/r regimen they are currently on)
* Patient's viral load have not been consistently <50 copies per ml for 6 months or longer.
* Patients initiated lipid lowering agents during the preceding 3 months
* Patients with any medical disorder or history of any illness which, in the opinion of the investigator, that the use of study medications is contraindicated or might confound the results of the study or pose additional risk in administering study drugs to the patient
* Pregnant, wish to become pregnant during the study period or breastfeeding women
* Patients who are lack of expectation to maintain assigned study medication during study period
* Patients who have received therapy with investigational drugs in the previous 3 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The proportion of patient-reported clinical adverse events | Week 4, 12-16, 28-32, 48
  The proportion of patient-reported clinical adverse events in total and by severity (based on symptom distress module) at 4 weeks, The proportion of patient-reported clinical adverse events in total and by severity (based on symptom distress module) at 12-16 weeks, The proportion of patient-reported clinical adverse events in total and by severity (based on symptom distress module) at 28-32 weeks, The proportion of patient-reported clinical adverse events in total and by severity (based on symptom distress module) at 48 weeks

SECONDARY OUTCOMES:
The proportion of patients who are free of "virological failure" | Week 4, 12-16, 28-32, 48
  The proportion of patients who are free of "virological failure" at week 4 after switch, The proportion of patients who are free of "virological failure" at week 12-16 after switch, The proportion of patients who are free of "virological failure" at week 28-32 after switch, The proportion of patients who are free of "virological failure" at week 48 after switch
The change from baseline in CD4 cell counts | Week 4, 12-16, 28-32, 48
  The change from baseline in CD4 cell counts at week 4 after switch, The change from baseline in CD4 cell counts at week 12-16 after switch, The change from baseline in CD4 cell counts at week 28-32 after switch, The change from baseline in CD4 cell counts at week 48 after switch
the change from baseline in life quality (based on the MOS-HIV questionnaire) | week 12-16, 48
  The change from baseline in quality of life (based on the MOS-HIV questionnaire) at week 12-16 after switch, The change from baseline in quality of life (based on the MOS-HIV questionnaire) at week 48 after switch.
The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) | Week 4, 12-16, 28-32, 48
  The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) at 4 weeks, The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) at 12-16 weeks, The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) at 28-32 weeks, The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) at 48 weeks
The proportion of patients with treatment failure | Week 4, 12-16, 28-32, 48
  The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) at 4 weeks, The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) at 12-16 weeks, The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) at 28-32 weeks, The percent changes from baseline in plasma lipid profiles (total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides) at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hsi-Hsun Lin, MD, Principal Investigator — E-DA Hospital
Locations (7):
- Taiwan (7):
  - E-Da Hospital, Kaohsiung, Taiwan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei City Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walensky RP. The survival benefits of AIDS treatment in the US. J Infect Dis 2006;194:11-19 Lennox JL. Safety and efficacy of raltegravir-based versus efavirenz-based combination therapy in treatment-naive patients with HIV-1 infection. Lancet 2009;374:796-806 Steigbigel RT. Long-term efficacy and safety of Raltegravir combined with optimized background therapy in treatment-experienced patients with drug-resistant HIV infection. Clin Infect Dis 2010;50:605-12 Eron JJ. Switch to raltegravir-based regimen versus continuation of a lopinavir-ritonavir-based regimen in stable HIV-infected patients with suppressed viraemia (SWITCHMRK 1 and 2). Lancet 2010;375:396-407 Martinex E. Substitution of raltegravir for ritonavir-boosted protease inhibitors in HIV-infected patients: the SPIRAL study. AIDS 2010, 24:1697-1707 Division of AIDS(DAIDS). Toxicity guideline for adults. http://rcc.tech-res.com/safetyand pharmacovigilance(accessed Apr 15, 2011)